CLINICAL TRIAL: NCT06521385
Title: Comparison of Non-invasive Respiratory Monitoring System (RMS) to Capnography for Respiratory Rate (RR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makani Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Makani-004
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Device Arm (Experimental): Subjects with both the reference and experimental device placed for paired data collection
  Interventions: Device: Makani Science Respiratory Monitoring System

INTERVENTIONS:
Device: Makani Science Respiratory Monitoring System — Subjects monitored by the Makani Science Respiratory Monitoring System

SUMMARY:
The goal of this clinical trial is to compare the performance of a novel non-invasive respiratory monitoring system against the gold standard methods (capnography) in human subjects. The main question it aims to answer is whether the novel monitoring system comparable to the current standards.

ELIGIBILITY:
Inclusion Criteria:

* Between age of 22-99
* BMI between 15 and 40 kg/m^2

Exclusion Criteria:

* Medical history of serious symptomatic, cardiac, or pulmonary disease.
* History of serious skin irritation (severe rash or blisters) caused by medical adhesives (tape).
* Cannot lay still for one (1) hour.
* Cannot give written informed consent.
* Unable to follow instructions.

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate Accuracy Compared Between Experimental and Reference Devices | 1 hour
  Accuracy (mean absolute error) of the subject respiratory rate (breaths/minute) measured by the Makani Science system (experimental device) compared against respiratory rate measured by capnography (reference device) for minute long segments.

SECONDARY OUTCOMES:
Respiratory Rate Bias Compared Between Experimental and Reference Devices | 1 hour
  Bias of the subject respiratory rate (breaths/minute) measured by the Makani Science system (experimental device) compared against respiratory rate measured by capnography (reference device) for minute long segments.
Makani Science System Performance after Simulated Breathing Artifacts | 15 minutes
  Accuracy (mean absolute error) of the subject respiratory rate (breaths/minute) measured by the Makani Science system (experimental device) compared against respiratory rate measured by capnography (reference device) after subject performed simulated breathing maneuvers.
Makani Science System Performance after Position Change | 15 minutes
  Accuracy (mean absolute error) of the subject respiratory rate (breaths/minute) measured by the Makani Science system (experimental device) compared against respiratory rate measured by capnography (reference device) after the subject shifts position.

CONTACTS AND LOCATIONS:
Locations (1):
- Illumination Foundation, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No